CLINICAL TRIAL: NCT04069845
Title: A Registry Study on the Risk Factors of Interstitial Pneumonia in Lymphoma Patients Treated With Liposomal Doxorubicin
Brief Title: A Registry Study in Lymphoma Patients Treated With Liposomal Doxorubicin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, professor, Ruijin Hospital
Other Study IDs: Realipo-01
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — liposomal doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liposomal doxorubicin treatment: intravenous liposomal doxorubicin
  Interventions: Drug: liposomal doxorubicin

INTERVENTIONS:
Drug: liposomal doxorubicin — intravenous liposomal doxorubicin

SUMMARY:
This study is to evaluate the incidence of interstitial pneumonia in lymphoma patients treated with liposomal doxorubucin. The treatment response and other adverse events will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed lymphoma
* 18-80 years
* ECOG<= 2
* newly diagnosed lymphoma
* liposomal doxorubicin is planned in the treatment
* normal lung function
* no history or malignancy
* informed consented

Exclusion Criteria:

* history of malignancy, now in the treatment
* pregnant
* serious infection
* other uncontrollable conditions judged by the investigator

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: de novo lymphoma patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of interstitial pneumonia | up to one month after completion of study treatment
  interstitial pneumonia is defined as positive CT scan with or without positive respiratory symptoms

SECONDARY OUTCOMES:
overall response rate | 21 days after completion of study treatment
  percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria
adverse events | up to 30 days after completion of study treatment
  number of participants with treatment-related adverse events mainly include liposomal related AEs, eg cardiotoxicity and the incidence of hand-foot syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No